CLINICAL TRIAL: NCT03065036
Title: A Prospective, Multi-Center Evaluation of the Hydrus Aqueous Implant (Standard and Low-Profile) for Lowering Intraocular Pressure (IOP) in Subjects With Mild to Advanced Primary Open Angle Glaucoma (POAG) With or Without a Cataract
Brief Title: Safety and Efficacy Study of the Hydrus Aqueous Implant in Subjects With POAG
Acronym: POAG
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ivantis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-09-001; HYDRUS I (Other: Germany: Federal Institute for Drugs and Medical Devices)
Record Dates: First submitted 2012-02-29; First posted 2017-02-27 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Primary Open Angle Glaucoma
Keywords: Primary Open Angle Glaucoma; POAG
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydrus Aqueous Implant (Experimental): Hydrus implanted into Schlemm's Canal.
  Interventions: Drug: prestudy topical glaucoma medications
- IOL placement and Hydrus implant (Other): Cataract Extraction with IOL placement and Hydrus implant into Schlemm's canal
  Interventions: Drug: prestudy topical glaucoma medications

INTERVENTIONS:
Drug: prestudy topical glaucoma medications — Reintroduction of prestudy topical glaucoma medications, introduced one medication at a time during each study visit, as necessary.

SUMMARY:
The purpose of this study is to evaluate the ocular hypotensive effect of the Hydrus Aqueous Implant (Standard and Low-Profile), as determined by the change in IOP from baseline (preoperative) and change in the number of glaucoma medications from baseline.

DETAILED DESCRIPTION:
This is a prospective, multi-center study that will examine subjects with documented mild to advanced primary open angle glaucoma (POAG), who may or may not have a cataract requiring removal and placement of an intraocular lens.

Study subjects will be grouped by the severity of their disease (either mild/moderate or advanced). If all inclusion and exclusion criteria are met subjects in all four groups will be implanted with the Hydrus Aqueous Implant. Subjects in whom a cataract is present will undergo standard cataract removal and IOL implantation concurrent with implantation of the Hydrus.

Postoperatively, subjects will undergo a complete ophthalmic evaluation at regularly scheduled intervals.

ELIGIBILITY:
Inclusion Criteria:

* Elevated intraocular pressure (IOP)
* Diagnosis of mild to advanced open-angle glaucoma
* Shaffer Grade III
* Mental capacity to cooperate when undergoing operative and postoperative examination
* 18 years of age or older
* Provide written informed consent
* Willing and able to return to scheduled follow-up examinations for 24-months

Exclusion Criteria:

* Closed-angle and narrow-angle forms of glaucoma
* Secondary glaucomas
* Congenital or developmental glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change in IOP of study eye between each randomized group | Baseline & One year
  Effectiveness will be determined by comparing the IOP at the baseline (pre-operative) visit to the the IOP at the 12 month post-operative visit.

SECONDARY OUTCOMES:
Change in glaucoma medications | Baseline & One year
  Calculate the change in the number of glaucoma medications from baseline (pre-operative) visit to the 12-month post-operative visit.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Manfred Tetz, MD, Principal Investigator — Augentagesklinik Spreebogen Berlin
Locations (5):
- University Medical Center Vienna, Vienna, Austria
- Germany (3):
  - Aurelios Augenzentrum, Recklinghausen, Erlbruch
  - Berlin
  - Universitatsmedizin der Johannes Gutenberg-Universitat Mainz Augenklinik und Poliklinik, Mainz
- Tijuana, Estado de Baja California, Mexico

IPD SHARING:
Plan to Share IPD: No